CLINICAL TRIAL: NCT06619925
Title: A Cohort Study of After-school Exercise Services in Promoting Myopia and Physical and Mental Health in Children
Brief Title: The Role of After-school Exercise Services in Promoting Myopia and Physical and Mental Health in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor, Anhui Medical University
Organization: Anhui Medical University (Other)
Other Study IDs: 20240909
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Common Diseases; Joint Prevention; Students; After-school Extended Sports Service
Keywords: common diseases; joint prevention; after-school extended sports service

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- after-school extended sports service: Impact of voluntary participation in different types (e.g. outdoor physical activities, indoor physical activities, ball games, calisthenics, etc.), intensity and duration of after-school extended physical education services on children's myopia and other physical and psychological well-being
  Interventions: Behavioral: after-school extended sports service
- non-after school extended sports service: Students in the same grade as the exposure group but participating in after-school non-physical education extended services (e.g., homework help, static activities such as calligraphy, chess, etc.) served as a control group, aiming to maximise the control of the influence of potential factors other than physical activity on the results of the study.
  Interventions: Behavioral: non-after school extended sports service

INTERVENTIONS:
Behavioral: after-school extended sports service — Impact of voluntary participation in different types (e.g. outdoor physical activities, indoor physical activities, ball games, calisthenics, etc.), intensity and duration of after-school extended physical education services on children's myopia and other physical and psychological well-being
  Groups: after-school extended sports service
Behavioral: non-after school extended sports service — Students in the same grade as the exposure group but participating in after-school non-physical education extended services (e.g., homework help, static activities such as calligraphy, chess, etc.) served as a control group, aiming to maximise the control of the influence of potential factors other than physical activity on the results of the study.
  Groups: non-after school extended sports service

SUMMARY:
This project is a prospective cohort study to evaluate the impact of after-school extended physical education services on the visual health, physical health indicators, and mental health of children and adolescents participating in these services over a one-year period. The study collected data on the participation rate, duration, activity content, and organisational form of the after-school extended hours service through a questionnaire; the demographic characteristics, sleeping habits, and dietary habits of the participants through a self-administered questionnaire on the multidisease behaviour of children and adolescents; the intensity of the activities of the students who participated in the after-school extended hours service was investigated through an accelerometer and a physical activity questionnaire; and data on students' visual acuity, body mass index, and mental health status were collected through a medical check-up. Students' visual acuity data, body mass index, maximum oxygen uptake, and other indicators of physical health and mental health were collected through physical examination, and data on changes in one year were collected through half-yearly/follow-up visits to establish a cohort to evaluate the effects of after-school extended hours services on students' myopia rates, physical health and mental health levels by different types, intensity and duration of exercise.

DETAILED DESCRIPTION:
Students in grades 1-6 of several primary schools were selected as the study subjects. According to the baseline survey, the study subjects were divided into after-school extended physical education service group and non-after-school extended physical education service group, and their behavioural habits as well as the contents of the after-school extended physical education service, visual acuity, BMI, cardiorespiratory fitness, spinal curvature abnormality, and mental health were investigated by means of questionnaires and other tools, so as to analyse the relationship between after-school extended physical education service and the physical and mental health of the students.

ELIGIBILITY:
Inclusion Criteria:

* ① Those who voluntarily participate in the after-school extended hours service;

  * Those who voluntarily participate in this study and sign the informed consent; ③ Basic reading, writing and comprehension skills to understand the questionnaire and be able to answer it;

Exclusion Criteria:

* ① Unfit to participate in sports activities for health or physical reasons; ② Suffering from glaucoma, glaucoma and other diseases.

  * Those who suffer from glaucoma, strabismus, refractive error and other eye diseases that affect vision;

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Students in grades 1-6 in a number of primary schools in a city were selected for the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
body mass index | At baseline, month 6 and month 12
  Among school-age children (5-9 years) and adolescents (10-19 years), BMI to determine whether they are obese or underweight depends on age and gender. Referring to the 2014 National Physical Fitness Standards for Students cut-off values were classified as normal, low weight, overweight, and obese.
cardiorespiratory fitness | At baseline, month 6 and month 12
  Cardiorespiratory endurance in children and adolescents was measured using the 20 m shutle run test.Extrapolated maximal oxygen uptake in children and adolescents using a 20 m round trip run = 62.103 + (0.302*Number of 20 mSRTs) - (0.877*BMI) - (4.874*Sex) - (0.465*Age) (M=0, F=1)
Spinal curvature abnormalities | At baseline, month 6 and month 12
  Referring to the standard 'Primary screening of spinal curvature abnormalities in children and adolescents' (GB/T 16133-2014), the visual inspection method, the forward bending test (FBT), and the angle of trunk rotation measurement (ATR), and the combination of the three methods were used to carry out the screening of spinal curvature abnormalities in children and adolescents. The type of scoliosis was assessed according to the combination of the three tests, and was classified as no scoliosis, scoliosis I degree, scoliosis II degree, and scoliosis III degree.
mental health | At baseline, month 6 and month 12
  Mental health status was measured using the Strengths and Difficulties Questionnaire (SDQ) (Chinese version) , which consists of 25 questions with five dimensions: emotional problems, peer relationships, conduct problems, hyperactivity/attention problems and pro-social behaviour. Each question was assigned a score of 0-2 according to 'does not meet', 'somewhat meets' and 'fully meets', with some of the entries reversed; the total score for all questions was calculated, with a range of 0-40, with higher scores representing closer to abnormality.
myopic | At baseline, month 6 and month 12
  Screening myopia was defined as SE≤-0.50D determined by computerised optometry under non-ciliary muscle paralysis when children and adolescents aged 6 years or older had a UCVA < 5.0; mild myopia: -3.00D< SE≤-0.50D; moderate myopia: -6.00D <SE≤﹣3.00D; high myopia: SE ≤ -6.00 D. Myopia progression was defined as myopia progression if the study subjects baseline myopia progressed to more severe myopia at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Cao Cai yun, Principal Investigator — Anhui Medical University

IPD SHARING:
Plan to Share IPD: No